CLINICAL TRIAL: NCT06020586
Title: Phase 2 Study to Evaluate the Efficacy and Safety of ECOHAIR Hair Lotion in the Accelerated Recovery of Chemotherapy-induced Alopecia.
Brief Title: Study To Evaluate The Efficacy And Safety Profile of ECOHAIR in Chemo-induced Alopecia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oncología Ángel H. Roffo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: roffo
Record Dates: First submitted 2023-06-01; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Chemotherapy-induced Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hair lotion (Experimental)
  Interventions: Other: hair lotion

INTERVENTIONS:
Other: hair lotion — ECOHAIR

SUMMARY:
This is a Phase 2, single-center study designed to determine the effect of ECOHAIR topical solution on scalp hair growth evaluated objectively ( images) and subjectively ( patient and investigator reports). A total of 22 subjects are planned to be enrolled, 15 in a prospective single-arm phase in which they will receive the study treatment and 7 controls. Patients should have a clinical diagnosis of chemotherapy-induced alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with stage I to III breast/ovarian cancer aged 18 to 65 years.
* Receiving chemotherapeutic agents containing taxanes and/or anthracyclines.
* Willing to agree to shave thinning hair at baseline.
* Willingness to be photographed and consent to photographic disclosure.
* Able to understand and willing to sign an informed consent form.
* Willing and able to follow all study instructions and attend all study visits.
* Subjects taking thyroid replacement medication must be on stable doses for 6 months prior to enrollment and remain on the same maintenance dose throughout the study.
* If female of childbearing age, must have a negative serum or urine pregnancy test at screnning (visit 0). Use a highly effective method of contraception during the study; do not plan a pregnancy for the duration of the study.

Exclusion Criteria:

* Use of any products or devices used to promote scalp hair growth (e.g., finasteride or minoxidil, L-tyrosine, cold caps).
* Sensitivity or allergy to any ingredient in the Ecohair product.
* Active skin disease on the scalp (such as psoriasis or seborrheic dermatitis) or history of skin disease on the scalp that, in the opinion of the investigator, may interfere with the efficacy or safety evaluations of the study.
* Active scalp trauma or other condition affecting the scalp that, in the opinion of the investigator may interfere with the conduct of the study or evaluations.
* The presence of a permanent or difficult to remove hairpiece or wig that, in the opinion of the investigator, will interfere with study evaluations if not removed at each visit.
* Failure to be able to perform assigned clinical visits.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of scalp surface area covered at 30 days. | 30 days
  The primary efficacy assessment is hair count in the target area (in a 1 cm2
  circular area) using trichoscopy imaging.
Time to event, defined as the time from the start of treatment to achieve 100% total hair coverage of the scalp. | baseline-30 days

SECONDARY OUTCOMES:
Scalp hair density at 30 days. | 30 days
Subject satisfaction questionnare. | baseline-30 days
  questionnaire is related to satisfaction with the outcome of the treatment (lotion).
Incidence and severity of local skin reactions. severity according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0) | baseline- 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Roffo, Caba, Buenos Aires, Argentina